CLINICAL TRIAL: NCT02651662
Title: A Phase 1 Study to Assess Safety and Tolerability of Odronextamab (REGN1979) an Anti-CD20 x Anti-CD3 Bispecific Monoclonal Antibody, and Cemiplimab (REGN2810), an Anti-Programmed Death-1 Monoclonal Antibody in Patients With B-Cell Malignancies (CLIO-1)
Brief Title: A Study to Learn How Safe and Tolerable Odronextamab and Cemiplimab Are in Adult Patients With B-cell Malignancies
Acronym: CLIO-1
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R1979-ONC-1504; 2015-001697-17 (EudraCT Number); 2023-508209-25-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2016-01-05; First posted 2016-01-11 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory Aggressive B-Cell Lymphoma
Keywords: B-Cell Non-Hodgkin Lymphoma (B-NHL)
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation phase (Experimental): Safety assessment of odronextamab in combination with cemiplimab and selection of recommended phase 2 dose (RP2D) regimen(s) for the combination of odronextamab and cemiplimab.
  Interventions: Drug: cemiplimab; Drug: odronextamab
- Dose expansion phase (Experimental): RP2D administration of the combination treatment.
  Interventions: Drug: cemiplimab; Drug: odronextamab

INTERVENTIONS:
Drug: cemiplimab — Administration via intravenous (IV) infusion. The dose(s) received will be according to dose level (DL) cohort assignment, as described in the protocol.
  Other Names: REGN2810; Libtayo
Drug: odronextamab — Administration IV infusion. The dose(s) received will be according to DL cohort assignment, as described in the protocol.
  Other Names: REGN1979

SUMMARY:
This study is researching a combination of 2 experimental drugs, referred to as "study drugs", called odronextamab (also known as REGN1979) and cemiplimab (also known as REGN2810). The study is focused on patients who have relapse/refractory aggressive B-cell lymphoma. The aim of the study is to see how safe and tolerable the study drugs are, and to define the recommended dose regimen for the combination with odronextamab.

This study is also looking at several other research questions, including:

* What side effects may happen from taking the study drugs
* How effective the study drugs are against the disease
* How much study drug is in the blood at different times
* Whether the body makes substances or protein called antibodies against the study drugs (that could make the drugs less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Have documented CD20+ aggressive B-cell NHL that is either not responsive to or relapsed after at least 2 prior lines of systemic therapy, for whom treatment with an anti-CD20 antibody may be appropriate. In addition, prior treatments should at least contain an anti-CD20 antibody and an alkylating agent.
2. Must have at least 1 nodal lesion (≥1.5 cm), or at least one extranodal lesion with longest transverse diameter (LDi) greater than 1.0 cm, documented by diagnostic imaging (computed tomography [CT] or magnetic resonance imaging [MRI]).
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
4. Adequate bone marrow and hepatic function, as defined in the protocol
5. Willing and able to comply with clinic visits and study-related procedures
6. Provide signed informed consent

Key Exclusion Criteria:

1. Primary central nervous system (CNS) lymphoma, or known or suspected CNS involvement by non-primary CNS NHL
2. History of or current relevant CNS pathology, as described in the protocol
3. Ongoing or recent (within 2 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments, which may suggest risk for immune-mediated adverse events (iAEs)
4. Prior therapies, as described in the protocol
5. Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection or other uncontrolled infection
6. Cytomegalovirus infection as noted by detectable levels on peripheral blood polymerase chain reaction (PCR) assay until the infection is well controlled.
7. Known hypersensitivity to both allopurinol and rasburicase
8. Pregnant or breastfeeding women
9. Women of childbearing potential, or men who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 6 months after the last dose, as defined in the protocol
10. Patients prior diagnosis of hemophagocytic lymphohistiocytosis (HLH) or macrophage activation syndrome (MAS)

Note: Other protocol-defined Inclusion/Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) of cemiplimab in combination with odronextamab | Up to 28 days
Incidence of treatment emergent adverse events (TEAEs) of cemiplimab in combination with odronextamab | Up to 18 months
Severity of TEAEs of cemiplimab in combination with odronextamab | Up to 18 months
Incidence of adverse events of special interest (AESIs) of cemiplimab in combination with odronextamab | Up to 18 months
Severity of AESIs of cemiplimab in combination with odronextamab | Up to 18 months

SECONDARY OUTCOMES:
Odronextamab and cemiplimab concentrations in serum | Up to 18 months
Incidence of anti-drug antibodies (ADAs) to odronextamab and cemiplimab over time | Up to 18 months
Titer of ADAs to odronextamab and cemiplimab over time | Up to 18 months
Incidence of neutralizing antibodies (Nabs) to odronextamab and cemiplimab over time | Up to 18 months
Titer of Nabs to odronextamab and cemiplimab over time | Up to 18 months
Overall response rate as assessed by investigator | Up to 18 months
Complete response (CR) rate as assessed by investigator | Up to 18 months
Duration of response as assessed by investigator | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (30):
- United States (5):
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber/Harvard Cancer Center - PO box 849168, Boston, Massachusetts
  - Harvard Medical School - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
- Austria (2):
  - Uniklinikum Salzburg (LKH) Universitatsklinik fur Innere Medizin III, Salzburg
  - Medical University Vienna, Vienna
- Germany (3):
  - University Hospital Frankfurt, Frankfurt am Main
  - Universitatsklinikum Jena, Jena
  - Universitatsklinikum Schleswig-Holstein, Campus Kiel, Kiel
- Israel (4):
  - Soroka, Beersheba
  - Hadassah Medical Center, Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Poland (5):
  - Pratia MCM Krakow, Krakow, Malopolska
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Pratia Onkologia Katowice, Katowice
  - Copernicus Memorial Hospital, Lodz
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy Warszawa, Warsaw
- Spain (11):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Institut Catala dOncologia (ICO Hospitalet), Barcelona
  - MD Anderson Cancer Center- Madrid, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/